CLINICAL TRIAL: NCT01606787
Title: Phase 3 Trial of Intravenous Mannitol Use During Partial Nephrectomy Prior to Renal Ischemia and Impact on Renal Function Outcomes
Brief Title: Mannitol Use During Partial Nephrectomy Prior to Renal Ischemia and Impact on Renal Function Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-079
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-02

CONDITIONS: Renal Cancer
Keywords: Kidney; MANNITOL; PLACEBO; Partial Nephrectomy; 12-079
MeSH Terms: conditions — Kidney Neoplasms | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- mannitol arm (Experimental): This study is a prospective randomized double blind placebo controlled trial comparing renal function outcomes in patients undergoing partial nephrectomy for renal tumors. Patients will be randomized in 1:1 fashion to receive mannitol or saline provided intravenously within 30 minutes prior to renal vascular clamping for performing partial nephrectomy.
  Interventions: Drug: mannitol
- placebo arm (Placebo Comparator): This study is a prospective randomized double blind placebo controlled trial comparing renal function outcomes in patients undergoing partial nephrectomy for renal tumors. Patients will be randomized in 1:1 fashion to receive mannitol or saline provided intravenously within 30 minutes prior to renal vascular clamping for performing partial nephrectomy.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: mannitol — After induction of general anesthesia Normosol or Lactated Ringers , at a target infusion rate of 10cc/kg (+/- 1cc/kg), will be administered over the first hour of surgery. After the first hour of surgery IV fluid will be administered at 6cc/kg (+/- 1cc/kg) intended to maintain a minimum systolic blood pressure of 90-100mmHg and a minimum urine output of 0.5cc/kg/hour. The treatment arm will receive a standard dose of 12.5 grams of mannitol (200 cc of a 6.25% mannitol solution) intravenously completely infused through an existing intravenous access catheter within 30 minutes prior to renal artery clamping.
  Arms: mannitol arm
Other: placebo — After induction of general anesthesia Normosol or Lactated Ringers at a target infusion rate of 10cc/kg (+/- 1cc/kg), will be administered over the first hour of surgery. After the first hour of surgery IV fluid will be administered at 6cc/kg (+/- 1cc/kg) intended to maintain a minimum systolic blood pressure of 90-100mmHg and a minimum urine output of 0.5cc/kg/hour. The placebo arm will receive 200cc of normal saline completely infused within 30 minutes prior to renal artery clamping.
  Arms: placebo arm

SUMMARY:
The purpose of this study is to determine if a medication called mannitol, can help the kidney maintain its function after kidney surgery. Mannitol is used to cause an increase in urine production (it is a diuretic). For many years, mannitol has been given to patients in the hope it would improve the kidney's circulation, and in doing so reduce the impact of the surgery on the kidney.

Mannitol is given during the surgery before the blood supply to the kidney is stopped. The blood supply to the kidney is stopped in order to minimize any blood loss during the removal of the tumor, and also to assist the surgeons view of the kidney anatomy. Once the tumor is removed the blood supply to the kidney is resumed. Sometimes a side effect of this temporary reduction in blood supply to the kidney is the loss of some kidney function. This may happen either in the short term (right away) or long term (months or years later). In studies done on animals, mannitol was able to lessen this damage to kidney function. However, no human study has ever confirmed that mannitol has the same helpful effect in humans. There is some suggestion that it may have no effect. Because sufficient research has yet to be done on humans, many surgeons do not give mannitol. A recent study, conducted at Memorial Sloan Kettering which looked back at patients who had undergone partial nephrectomies, an operation where only the portion of the kidney that contains the tumor is removed and enables the normal, unaffected portion of the kidney to be preserved. The results of this study demonstrated no significant difference in kidney function when the investigators compared patients who were given mannitol to those who were not. The investigators hope that this study will help clarify the effectiveness or not of mannitol on kidney function. During the surgery to remove the kidney tumor, patients will receive either mannitol or a placebo. A placebo, is a harmless medication that has no effects. The impact of mannitol compared to the placebo will be assessed by routine blood tests and imaging (kidney scan) 6 months after your surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = to 18 years
* Scheduled for partial nephrectomy at MSKCC (open or minimally invasive technique) during which renal ischemia is anticipated
* Preoperative eGFR > 45 cc/min/1.73m2 as measured by the CKD-EPI study equation

Exclusion Criteria:

* Allergy to mannitol
* Severe renal impairment (stage 3B) defined as eGFR < 45 cc/min/1.73m2 as measured by the CKD-EPI calculation.
* Combined major surgical cases that include a partial nephrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-05-22 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coleman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Spaliviero M, Power NE, Murray KS, Sjoberg DD, Benfante NE, Bernstein ML, Wren J, Russo P, Coleman JA. Intravenous Mannitol Versus Placebo During Partial Nephrectomy in Patients with Normal Kidney Function: A Double-blind, Clinically-integrated, Randomized Trial. Eur Urol. 2018 Jan;73(1):53-59. doi: 10.1016/j.eururo.2017.07.038. Epub 2017 Aug 16. PMID 28822586
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mannitol Arm | Placebo Arm
Started | 105 | 105
Completed | 101 | 98
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Surgery canceled | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mannitol Arm | Placebo Arm | Total
Number analyzed (Participants) | 101 | 98 | 199
Age, Continuous [Median (Full Range); unit: years] | 60 [50 to 66] | 56 [48 to 63] | 58 [48 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 65 | 61 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 10 | 15
  White | 81 | 80 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 3 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101 | 98 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to 6 Months
Description: The difference will be assessed with an ANCOVA model with eGFR 6 months after surgery (+/- 2 months) as the outcome and treatment group, surgical technique, and preoperative eGFR as covariates. We will report a two-tailed p-value and a 95% confidence interval for the difference between groups. If a patient does not have an eGFR measurement between 5-7 months after surgery and has both a measurement between 3-5 months and 7-12 months after surgery, then the 6 month eGFR measurement will be linearly interpolated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change from preoperative eGFR
Arm/Group | Mannitol Arm | Placebo Arm
Number analyzed (Participants) | 101 | 99
% change from preoperative eGFR | -8.5 (14) | -8.4 (12)

2. Secondary Outcome: Percent Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to 6 Weeks
Description: between treatment groups at 6 weeks (+/- 4 weeks) after surgery with postoperative eGFR as the outcome, and treatment group, surgical technique, and preoperative eGFR as covariates. We will also use the ANCOVA on the absolute level of eGFR because this has the greatest statistical power. However, the estimate produced by ANCOVA - a mean difference in eGFR levels - is of incomplete clinical interpretability.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: % change from preoperative eGFR
Arm/Group | Mannitol Arm | Placebo Arm
Number analyzed (Participants) | 101 | 99
% change from preoperative eGFR | -6.2 (13) | -9.4 (14)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Mannitol Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/101 | 2/98
Serious Adverse Events (participants affected / at risk) | 19/101 | 11/98
Other Adverse Events (participants affected / at risk) | 2/101 | 7/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mannitol Arm (N=101) | Placebo Arm (N=98)
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 2 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Hematoma (Vascular disorders) | 2 | 2
Hematuria (Renal and urinary disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Urinary Fistula (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Injury/poison & proced complications Other, spec (Injury, poisoning and procedural complications) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mannitol Arm (N=101) | Placebo Arm (N=98)
Urinary Fistula (Renal and urinary disorders) | 1 | 1
Fever (General disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Injury/poison & proced complications Other, spec (Injury, poisoning and procedural complications) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT01606787/Prot_SAP_000.pdf